CLINICAL TRIAL: NCT04687267
Title: Gestione Conservativa di Lesioni CIN2 e Valutazione di Biomarcatori Indicativi di Regressione
Brief Title: Conservative Management of CIN2 Lesions and Biomarkers Evaluation
Status: Completed | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Azienda ULSS 3 Serenissima (Other); Azienda Ulss 6 Euganea (Other); Azienda Ulss 2 Marca Trevigiana (Other); Azienda Ulss 9 Scaligera (Other Government); Regione Veneto (Other)
Responsible Party: Principal Investigator, Annarosa Del Mistro, Head of HPV laboratory, Istituto Oncologico Veneto IRCCS
Other Study IDs: CIN2-RSFR
Record Dates: First submitted 2020-12-10; First posted 2020-12-29 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: CIN2
Keywords: biomarkers; HPV; methylation; clinical outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical cells and DNA extracted therefrom to be used for biomarkers analyses, retained for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective study including women aged 25-45 years, adherent to the cervical screening program of four different centers of the Veneto region, with a diagnosis of CIN2 lesion. After enrollment according to predefined criteria, and informed consent to participate, the CIN2 lesions are managed by follow-up; cases with progressive lesions will be treated immediately, cases with CIN2 persistence for more than 12 months will be treated as well. Viral, molecular and immunocytochemical biomarkers will be studied, and evaluated in relation to the clinical outcome.

DETAILED DESCRIPTION:
Women aged 25-45 years, adherent to the organized population-based cervical screening program, with a histological diagnosis of CIN2 and fulfilling the inclusion criteria will be invited to participate to the study, previously providing specific information; in case of acceptance, informed consent is signed.

STUDY PROTOCOL:

The adherent women will attend periodical control visits:

* every 6 months up to 24 months, with performance of: pap test (PT) and colposcopy (with biopsy in case of visible alterations);
* at 6 and 12 months control visit: a liquid-based sample of cervical cells will be collected for the biomarkers' analyses.

BIOMARKERS:

1. - HPV search and partial HPV16/18 genotyping, by cobas 4800 high-risk HPV assay (Roche); PCR with MY09/MY11 consensus primers and full genotyping by restriction fragment length analysis, plus PCR with beta-globin primers (in-house);
2. - methylation analysis of the cellular genes FAM194A and hsa-mir124-2, by methylation-specific quantitative PCR test (qMSP - QIAsure methylation test, Qiagen);
3. - methylation analysis of the L1 and L2 viral genes of HPV types 16 and 18, by pyrosequencing;
4. - immunocytochemical analysis for p16INK4A/Ki67 proteins (dual stain), by p16INK4A/Ki67 immunocytochemical analysis by CINtec Plus kit (Roche).

ELIGIBILITY:
Inclusion Criteria:

* age range 25-45 years,
* CIN2 lesions located in the exocervix and completely visible at colposcopy.

Exclusion Criteria:

* age >45 years;
* history of previous high-grade lesions;
* squamo-columnar junction not completely visible (type 3);
* cytology with suspect or indicative for invasive lesion;
* lesions exclusively located in the endocervix;
* lesions located in the exocervix but not completely visible;
* pregnancy

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study is related to a disease of the female genital tract.
Study Population: Women attending organized population-based cervical cancer screening with a histological CIN2 lesion, meeting the selection criteria and consenting to participate.
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of spontaneous regression of CIN2 lesions | Through study completion, an average of 2 years.
  Eligible women will not be treated at diagnosis, but periodically followed-up. Treatment will be provided for progressive lesions and lesions persisting more than 12 months. The rates of lesion regression will be calculated: number of lesions regressed to CIN1 or normal / total number of cases.
CIN2 clinical outcome by HPV genotype | Through study completion, an average of 2 years.
  Rate of CIN2 regression will be calculated in relation to positivity for HPV16 vs positivity for other high-risk types (number of regressed HPV16-related CIN2 lesions / total number of HPV16-related CIN2 vs number of regressed non-HPV16-related CIN2 lesions / total number of non-HPV16-related CIN2 lesions).
CIN2 clinical outcome by DNA methylation | Through study completion, an average of 2 years.
  Rate of CIN2 regression will be calculated in relation to DNA methylation of cellular and viral genes (number of regressed hypermethylated CIN2 lesions / total number of CIN2 lesions with valid result for each gene analyzed).
CIN2 clinical outcome by p16/ki67 protein expression | Through study completion, an average of 2 years.
  Rate of CIN2 regression will be calculated in relation to positivity for p16/ki67 expression (number of regressed p16/ki67-positive CIN2 lesions / total number of CIN2 lesions with valid result for p16/ki67 expression).

SECONDARY OUTCOMES:
Adhesion to CIN2 conservative management. | 2 years
  The rate of eligible women consenting to participate to the study will be calculated (enrolled women / eligible women)

CONTACTS AND LOCATIONS:
Overall Officials: Tiziano Maggino, MD, Principal Investigator — Azienda ULSS 3 Serenissima
Locations (4):
- Italy (4):
  - Azienda ULSS 6 Euganea, Padua, PD
  - Azienda ULSS 2 Marca Trevigiana, Treviso, TV
  - Azienda ULSS 3 Serenissima, Mestre, VE
  - Azienda ULSS 9 Scaligera, Verona, VR

REFERENCES:
- [Background] Del Mistro A, Matteucci M, Insacco EA, Onnis G, Da Re F, Baboci L, Zorzi M, Minucci D. Long-Term Clinical Outcome after Treatment for High-Grade Cervical Lesions: A Retrospective Monoinstitutional Cohort Study. Biomed Res Int. 2015;2015:984528. doi: 10.1155/2015/984528. Epub 2015 Jun 9. PMID 26180819
- [Background] Del Mistro A, Frayle H, Rizzi M, Fantin G, Ferro A, Angeletti PM, Giorgi Rossi P, Altobelli E. Methylation analysis and HPV genotyping of self-collected cervical samples from women not responding to screening invitation and review of the literature. PLoS One. 2017 Mar 6;12(3):e0172226. doi: 10.1371/journal.pone.0172226. eCollection 2017. PMID 28263992
- [Background] Ordi J, Sagasta A, Munmany M, Rodriguez-Carunchio L, Torne A, del Pino M. Usefulness of p16/Ki67 immunostaining in the triage of women referred to colposcopy. Cancer Cytopathol. 2014 Mar;122(3):227-35. doi: 10.1002/cncy.21366. PMID 24757722
- [Background] Gillio-Tos A, Fiano V, Grasso C, Trevisan M, Gori S, Mongia A, De Marco L, Ronco G; New Technologies for Cervical Cancer Screening (NTCC) Working Group. Assessment of viral methylation levels for high risk HPV types by newly designed consensus primers PCR and pyrosequencing. PLoS One. 2018 Mar 26;13(3):e0194619. doi: 10.1371/journal.pone.0194619. eCollection 2018. PMID 29579066